CLINICAL TRIAL: NCT00205348
Title: Swallowing Function Before and After Surgery for Thyroid Goiter
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2002-093
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2017-08

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To date, there have been no comprehensive studies on swallowing function in patients undergoing surgery for multinodular goiter. We hypothesize that 1. Multinodular goiter has significant effect on swallowing function in symptomatic and asymptomatic patients, which can be demonstrated by a standardized questionnaire and a formal swallowing evaluation and 2. Surgery will improve swallowing function as measured post-operatively by these same parameters. Patients with multinodular goiter will be asked to fill out a validated survey (SWAL-QOL) on swallowing function in addition to undergoing a formal swallowing evaluation before and after surgery for multinodular goiter (subtotal thyroidectomy) and compared to patients undergoing total thyroidectomy for follicular cancer and less extensive thyroid surgery for other benign processes (lobectomy or lobectomy plus isthmusectomy).

DETAILED DESCRIPTION:
Detailed description not desired.

ELIGIBILITY:
Inclusion Criteria:

* thyroidectomy

Exclusion Criteria:

* na

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing thyroid surgery
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2002-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Chen, MD, Principal Investigator — University of Wisconsin Medical School

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing thyroid surgery from May 2002 to December 2004 completed the SWAL-QOL questionnaire before and one year after surgery.
Groups:
- SWAL-QOL Questionnaire: Patients undergoing thyroid surgery from May 2002 to December 2004 completed the Swallowing Quality Of Life (SWAL-QOL)questionnaire before and one year after surgery. The SWAL-QOL is a 44 item tool that asks patients to rate several factors about 10 quality-of-life concepts related to swallowing on a 5 point scale.
  Data were collected on demographic and clinicopathologic variables, and comparisons were made to determine the effect of surgery on patients' perceptions of swallowing function.
Period: Overall Study
Arm/Group | SWAL-QOL Questionnaire
Started | 146
Completed | 116
Not Completed | 30

BASELINE CHARACTERISTICS:
Arm/Group | SWAL-QOL Questionnaire
Number analyzed (Participants) | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 116
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 116

OUTCOME MEASURES:

1. Primary Outcome: Swallowing Quality of Life
Description: The swallowing quality of life (SWAL-QOL) validated outcomes assessment tool will be used before and one year after surgery to measure changes in swallowing-related QOL in patients undergoing thyroid surgery. The SWAL-QOL is a 44 item tool that asks patients to rate several factors about 10 quality-of-life concepts related to swallowing on a 5 point scale.Data were collected on demographic and clinicopathologic variables, and comparisons were made to determine the effect of surgery on patients' perceptions of swallowing function. A score of 0 represents the least favorable state, and 100 the most favorable. It has been validated and has favorable psychometric properties, including high internal-consistency reliability and reproducibility. The scales of the instrument differentiate patients with oropharyngeal dysphagia from normal swallowers and are sensitive to clinically-relevant differences in dysphagia severity in patients with medically and surgically treated conditions.
Time Frame: One year
Population: All data will be analyzed using standard statistical tools including student T-test and ANOVA.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- SWAL-QOL Questionnaire: Patients undergoing thyroid surgery from May 2002 to December 2004 completed the Swallowing Quality Of Life (SWAL-QOL)questionnaire before and one year after surgery. The SWAL-QOL is a 44 item tool that asks patients to rate several factors about 10 quality-of-life concepts related to swallowing on a 5 point scale.
  Data were collected on demographic and clinicopathologic variables, and comparisons were made to determine the effect of surgery on patients' perceptions of swallowing function. A score of 0 represents the least favorable state, and 100 the most favorable.
Arm/Group | SWAL-QOL Questionnaire
Number analyzed (Participants) | 116
units on a scale
  Burden Score Before Surgery | 84.6 [0 to 100]
  Burden Score After Surgery | 92.3 [0 to 100]
  Physical Score Before Surgery | 81.2 [19.6 to 100]
  Physical Score After Surgery | 87.1 [26.8 to 100]
  Mental Score Before Surgery | 87.0 [0 to 100]
  Mental Score After Surgery | 93.1 [10 to 100]
  Fear Score Before Surgery | 87.0 [12.5 to 100]
  Fear Score After Surgery | 92.9 [25 to 100]
  Eating Desire Score Before Surgery | 92.5 [0 to 100]
  Eating Desire Score After Surgery | 94.5 [25 to 100]
  Eating Duration Score Before Surgery | 86.2 [0 to 100]
  Eating Duration Score After Surgery | 88.4 [0 to 100]
  Food Selection Score Before Surgery | 88.5 [0 to 100]
  Food Selection Score After Surgery | 93.8 [25 to 100]
  Sleep Score Before Surgery | 65.0 [0 to 100]
  Sleep Score After Surgery | 73.6 [0 to 100]
  Fatigue Score Before Surgery | 63.4 [0 to 100]
  Fatigue Score After Surgery | 71.5 [0 to 100]
  Social Score Before Surgery | 94.4 [20 to 100]
  Social Score After Surgery | 95.6 [25 to 100]
  Communication Score Before Surgery | 88.9 [0 to 100]
  Communication Score After Surgery | 91.9 [25 to 100]
Statistical Analysis 1: Comparison: SWAL-QOL Questionnaire; The statistical significance of the difference between pre-and post-operative scores for Burden was tested with the Wilcoxon signed-rank test; Test type: Superiority or Other; p = 0.0007, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: SWAL-QOL Questionnaire; The statistical significance of the difference between pre-and post-operative scores for Physical was tested with the Wilcoxon signed-rank test; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: SWAL-QOL Questionnaire; The statistical significance of the difference between pre-and post-operative scores for Mental was tested with the Wilcoxon signed-rank test; Test type: Superiority or Other; p = 0.0002, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: SWAL-QOL Questionnaire; The statistical significance of the difference between pre-and post-operative scores for Fear was tested with the Wilcoxon signed-rank test; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: SWAL-QOL Questionnaire; The statistical significance of the difference between pre-and post-operative scores for Eating Desire was tested with the Wilcoxon signed-rank test; Test type: Superiority or Other; p = 0.0973, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: SWAL-QOL Questionnaire; The statistical significance of the difference between pre-and post-operative scores for Eating Duration was tested with the Wilcoxon signed-rank test; Test type: Superiority or Other; p = 0.1772, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: SWAL-QOL Questionnaire; The statistical significance of the difference between pre-and post-operative scores for Food Selection was tested with the Wilcoxon signed-rank test; Test type: Superiority or Other; p = 0.0062, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: SWAL-QOL Questionnaire; The statistical significance of the difference between pre-and post-operative scores for Sleep was tested with the Wilcoxon signed-rank test; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: SWAL-QOL Questionnaire; The statistical significance of the difference between pre-and post-operative scores for Fatigue was tested with the Wilcoxon signed-rank test; Test type: Superiority or Other; p = 0.0002, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: SWAL-QOL Questionnaire; The statistical significance of the difference between pre-and post-operative scores for Social was tested with the Wilcoxon signed-rank test; Test type: Superiority or Other; p = 0.2125, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: SWAL-QOL Questionnaire; The statistical significance of the difference between pre-and post-operative scores for Communication was tested with the Wilcoxon signed-rank test; Test type: Superiority or Other; p = 0.0332, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | SWAL-QOL Questionnaire
Serious Adverse Events (participants affected / at risk) | 0/116
Other Adverse Events (participants affected / at risk) | 0/116

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No